CLINICAL TRIAL: NCT04743258
Title: Evaluation of Treatment Changes in Class II Div 1 Malocclusion With Bilateral Extraction of Maxillary First Premolars vs Full Arch Distalization: A Randomised Clinical Trial
Brief Title: Bilateral Premolar Extraction vs Distalization: A Randomised Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SONAL SURJEET
Record Dates: First submitted 2020-08-18; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXTRACTION (Experimental): treatment of class II div 1 malocclusion with bilateral maxillary premolar extraction
  Interventions: Procedure: MAXILLARY PREMOLAR EXTRACTION
- DISTALIZATION (Experimental): treatment of class II div 1 malocclusion with distalization using zygomatic miniplates
  Interventions: Procedure: DISTALIZATION

INTERVENTIONS:
Procedure: MAXILLARY PREMOLAR EXTRACTION — Patients will undergo bilateral maxillary 1st premolar extraction before bonding followed by leveling & alignment.
  Arms: EXTRACTION
Procedure: DISTALIZATION — Maxillary arch will be distalized with the help Zygomatic miniplates will be placed bilaterally.
  Arms: DISTALIZATION

SUMMARY:
Rationale: Class II Division 1 malocclusion is characterized by upper anterior teeth protrusion resulting in upper lip protrusion and convex facial profile, which are considered esthetically unfavorable. Treatment of class II malocclusion due to maxillary protrusion can be done with bilateral maxillary first premolar extraction followed by en-masse retraction of upper anterior teeth using mini implants placed between maxillary 2nd premolar & 1st molar.

Treatment of class II malocclusion due to maxillary protrusion without premolar extraction frequently requires distalization of maxillary molars into Class I molar relation by means of extra-oral or intraoral forces. Absolute skeletal anchorage, available 24 hours a day is an alternative method for molar distalization. Zygomatic miniplates fixed at a distance from the root apices, allows distalization of entire dentition as there is no interference between the fixation device and roots of the teeth.

Aims and Objectives: To evaluate dental, skeletal & soft tissue changes achieved with maxillary premolar extraction vs full arch distalization.

Method of study: Patients will be allocated randomly to 2 groups-G1 and G2. Patients in G1 will undergo bilateral maxillary 1st premolar extraction before bonding followed by leveling & alignment. Maxillary arch will be stabilized with the help of 0.019"×0.025" stainless steel wire. Hooks will be soldered on archwire used for stabilizing dentition. Mini implants will be placed under local anaesthesia between maxillary 2nd premolar & 1st molar. Ni-Ti closed coil spring will be used to apply a force for en masse retraction of maxillary anterior teeth .

In G2, treatment will be initiated by bonding 0.022" slot MBT preadjusted edgewise appliance. Maxillary arch will be stabilized with the help of 0.019"×0.025" stainless steel wire. Zygomatic miniplates will be placed bilaterally. Hooks will be soldered on archwire used for stabilizing dentition. Ni-Ti closed coil spring will be used to apply a force .

DETAILED DESCRIPTION:
The present study is a prospective, non-pharmacological, single blind, randomized clinical study to evaluate the skeletal, dental and soft tissue changes with distalization of entire maxillary dentition using bilateral maxillary 1st premolar extraction in comparison with zygomatic miniplates in class II division 1 patients. The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopaedics, in conjunction with the Department of Oral and Maxillofacial Surgery, P.G.I.D.S., Pt. B.D.Sharma University of Health Sciences, Rohtak. The study will be carried out after the institutional approval obtained from the ethical committee.

SOURCE OF DATA The study sample consists of 34 subjects selected from the patients attending the regular OPD at the Department of Orthodontics and DentofacialOrthopaedics for orthodontic treatment.

INCLUSION CRITERIA

* Non growing patients
* Complete bilateral Class II molar relationship at pre-treatment
* All permanent teeth upto the second molars should be present
* No or minor crowding in the maxillary arch
* Horizontal to average growth pattern.

EXCLUSION CRITERIA

* Subjects with a history of fixed orthodontic treatment.
* Crossbite
* Vertical growth pattern
* Any systemic disease affecting bone and general growth
* Poor oral hygiene
* Cleft patients
* Patients who fail to follow up or undergo complete treatment TARGET SAMPLE SIZE
* A sample size of 15 per group for the present study was calculated to detect a clinical difference of 3.9 mm with effect size 0.86 at 95% power and 5% significance level. To compensate for 10% dropouts the final sample size was calculated to be 17 per group.

INFORMED CONSENT OF THE PATIENT AND AGREEMENT TO BE RANDOMIZED A valid, written informed consent of the patient or parent/ guardian and an agreement to be randomized will be obtained from the patient before registering the patient in this clinical study. Patient will be informed about all the theoretical risks and benefits of the intervention under test (Annexure I). The patient will be given 72 hours to discuss the study with his/her family and take the decision regarding participation in the study.

RANDOMIZATION & ALLOCATION CONCEALMENT Randomization will be done by a person not involved in the trial using computer generated randomization list. The study subjects will be blinded regarding intervention group.

INTERVENTION AND DESIGN OF STUDY The main intervention in this prospective clinical study is the extraction of bilateral maxillary first premolars before initial leveling and alignment with retraction of anterior teeth using mini implants in first group (G1) and is the placement of zygomatic miniplates after initial leveling and alignment of maxillary dental arch in second group(G2) . The study consists of 2 groups with equal allocation of subjects in each group:- Group 1 (G1):- In this group, bilateral maxillary 1st premolars will be extracted followed by Levelling & alignment with 0.022" MBT preadjusted edgewise appliance. Maxillary arch will be stabilized with the help of 0.019" × 0.025" stainless steel wire. Placement of Mini implants bilaterally between maxillary 2nd premolar & 1st molar under LA. Hooks will be soldered on archwire used for stabilizing dentition. Ni-Ti closed coil spring will be used to apply force . Regular follow up of the patient will be done and records including cephalograms and study models will be taken post 6 months of application of NiTi closed coil spring Group 2 (G2):- In this group treatment will be initiated with 0.022" MBT preadjusted edgewise appliance. Maxillary arch will be stabilized with the help of 0.019" × 0.025" stainless steel wire. After that, bilateral Maxillary third molar will be extracted, if present followed by placement of zygomatic miniplates bilaterally under LA.Hooks will be soldered on archwire used for stabilizing dentition. Ni-Ti closed coil spring will be used to apply force . Regular follow up of the patient will be done and records including cephalograms and study models will be taken post 6 months of application of NiTi closed coil spring DATA COLLECTION The investigator will record the patient's name, address and contact number and other relevant case history records (Annexure II) will be taken. Cephalometric radiographs will be recorded before treatment and after 6 months of application of NiTi closed coil spring for assessment of hard and soft tissue changes. The pretreatment and post 6 months of application of NiTi closed coil spring the cephalometric radiographs will be analyzed. The relevant values will be entered in a predesigned format. (Annexure III, IV). Soft tissue profile changes between pretreatment and post treatment will be assessed on lateral cephalogram and the raters- orthodontist, laypersons,patients,parents and general dentists will assess changes in facial appearance on a visual analog scale with profile photographs and comparison will be done between the two groups. Patient perception will be assessed using questionare rating by patient regarding various parameters at 1week, 2 weeks, 1 month and 6 months after the placement of zygomatic miniplate or extraction Quality of life will also be assessed using questionnaire rating by patient at pre-treatment, mid-treatment and post treatment. Occlusal status changes between pre and post treatment will be assessed using PAR index(peer assessment rating between 2 groups).

STATISTICAL ANALYSIS The data will be entered into Microsoft Excel and analyzed using SPSS 21(Statistical Package For Social Sciences) package for relevant statistical comparison. Results will be presented in the form of tables and graphs.

Descriptive statistics and inferential statistics will be used. Data will be checked for normality. In all the analysis, the level of significance will be set a 5 percent.

ELIGIBILITY:
Inclusion Criteria:

1. Non growing patients
2. Complete bilateral Class II molar relationship at pre-treatment
3. All permanent teeth upto the second molars should be present
4. No or minor crowding in the maxillary arch
5. Horizontal to average growth pattern.

Exclusion Criteria:

1. Subjects with a history of fixed orthodontic treatment.
2. Crossbite
3. Vertical growth pattern
4. Any systemic disease affecting bone and general growth
5. Poor oral hygiene
6. Cleft patients
7. Patients who fail to follow up or undergo complete treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
skeletal angular changes | 28 months
  SNA angle Pre & Post after space closure in group 1 & achieving Class I molar relation in group 2
Maxillary dentoalveolar changes | 28 months
  maxillary incisor to NA angle Pre & Post after space closure in group 1 & achieving Class I molar relation in group 2
Soft tissue changes | 34 months
  soft tissue profile changes after distalization evaluated on lateral cephalogram and the raters- orthodontist, laypersons,patients,parents and general dentists will assess changes in facial appearance on a visual analog scale with profile photographs
overjet & overbite measured in mm | 28 months
  Pre & Post after space closure in group 1 & achieving Class I molar relation in group 2

SECONDARY OUTCOMES:
mandibular plane angle | [Time Frame: 28 months]
  changes in mandibular plane angle after distalization with zygomatic miniplates & comparison with enmasse anterior retraction with mini implants
airway changes | [Time Frame: 28 months]
  Changes in the upper-airway size will be measured by using lateral cephalometric radiographs taken before and after distalization

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol